CLINICAL TRIAL: NCT03555162
Title: Cerebral Bases of Tool Use and Tool Evolution
Brief Title: Study of the Cerebral Bases of Tool Use and Tool Evolution
Acronym: TOOLBOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0121
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Tool; fMRI; neuroimaging; Evolution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tool Use (Other): The fMRI experimental conditions in this arm will allow us to study the activity of the brain when using tools. Here only the fMRI experimental session is necessary. Tasks proposed to the participants within the fMRI scanner will be related to tool use. They will have to solve mechanical problems, to judge the appropriateness of hand postures for using tools, and to judge if tools presented share the same context of use, the same functional goals, the same hand postures for using them.These experimental conditions related to the BOLD measures given by the fMRI technique will allow us to draw hypotheses on the neurocognitive mechanisms at work when we use tools.
  Interventions: Other: fMRI
- Tool Evolution (Other): The fMRI experimental conditions in this arm will allow us to study the activity of the brain when we improve tools. Here the fMRI experimental session will be complemented by a cognitive psychology experiment, where participants will be given a tool to improve. Tasks proposed to the participants within the fMRI scanner will be related to cognitive functions that could be implicated in improving tools : creativity, technical reasinoning, logic, empathy. The BOLD measures realted to these experimental condfitions will be related to the ability of the participant to improve a tool, through General Linear Modeling.
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — Imaging examination

SUMMARY:
Tool use is considered to be the hallmark of complex cognitive adaptations that humans have achieved trough evolution, that provides an adaptive advantage to the human species. Even if nonhuman species do use tools too, human tool use is much more complex and sophisticated. Besides, only humans can make their tools evolve by improving them. If Man has special abilities for tool use, it has to be grounded in a specific neuroanatomical substrate. Humans and nonhumans share a similar prehension system located within the superior parietal lobe and the intraparietal sulcus. However, there is a human specificity : the surpramarginal gyrus within the left inferior parietal lobe is unique to Man, and could play a central role in tool use and tool evolution.

This project aims to study the neural correlates of human tool use with functional Magnetic Resonance Imaging (fMRI), to precise the cognitive mechanisms through which humans are able to use tools. We also wish to study what are the cognitive abilities that allow us to make our tools evolve by improving them, and the neural correlates associated.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18 and 65 years old
* Having given an informed consent for the study
* Being right-handed
* Being registered with the French Social Security System

Exclusion Criteria:

* No signature on the consent form, including inability to read or write French.
* Neurologic or psychiatric illness, known or revealed durnig the inclusion visit
* Substance intake ( taking psychoactive medications or recreational drugs) on the day of the experiment
* Noise intolerance
* Minor person, pregnant or breastfeeding woman
* Persons under curatorship or deprived of civil rights or deprived of their freedom
* Unable to fill a questionnaire (severe cognitive troubles)
* Subjects must not have metallic or electronic implants in the body : pacemakers or pacemaker wires, open heart surgery, artificial heart valve, brain aneurysm surgery, middle ear implant, hearing aid, braces or extensive dental work, cataract surgery or lens implant, implanted mechanical or electrical device, or artificial limb or joint o foreign metallic objects in the body (bullets, BBs, pellets, schrapnel, or metalwork fragments) or current or past employment as machinists, welders or metal workers, tattoos near the head or neck regions, permanent makeup
* Claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
BOLD effect | 1 hour
  The measure will be the Blood Oxygenation Level Dependent measure (BOLD) as permitted with functional Magnetic Resonance Imaging. This BOLD level will be collected for every voxel in the imaged brain, and at regular time intervals (TR = 3") during the experimental session (about one hour). This is standard procedure for fMRI experiments.
  Functional magnetic resonance imaging measures brain activity by detecting changes associated with blood flow This technique relies on the fact that cerebral blood flow and neuronal activation are coupled. When an area of the brain is in use, blood flow to that region also increases. The primary form of fMRI uses the BOLD contrast in response to an experimental condition, allowing researchers to track changes in oxygen comsumption on the brain, and therefore brain activity. BOLD efefct is computed by assessing the different relaxation times (T1 and T2) in the brain, as T1 and T2 are different in function of regional cerebral blood flows.

SECONDARY OUTCOMES:
Ability to improve a tool | 20 minutes
  Participants will be given metal wires and asked to build a tower as high as possible. For this, they will be able to observe the previous participant to inspire themselves. The measure collected will be the height of the tower, compared to the height of the tower of the previous participant.

CONTACTS AND LOCATIONS:
Overall Officials: Yves ROSSETTI, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Laboratoire d'Etude des Mécanismes Cognitifs (EMC) -Université Lumière Lyon 2, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lesourd M, Osiurak F, Martin J, Hague S, Laroze M, Clement G, Medeiros de Bustos E, Fargeix G, Magnin E, Moulin T. Neurocognitive mechanisms underlying action tool knowledge tasks: specificity of tool-tool compared to hand-tool compatibility tasks. Commun Biol. 2025 Apr 3;8(1):552. doi: 10.1038/s42003-025-07923-1. PMID 40181134
- [Background] Osiurak F, Federico G, Fournel A, Gaujoux V, Lamberton F, Ibarrola D, Rossetti Y, Lesourd M. Shaping the physical world to our ends through the left PF technical-cognition area. Elife. 2025 Apr 17;13:RP94578. doi: 10.7554/eLife.94578. PMID 40243287
- [Background] Lesourd M, Reynaud E, Navarro J, Gaujoux V, Faye-Vedrines A, Alexandre B, Baumard J, Federico G, Lamberton F, Ibarrola D, Rossetti Y, Osiurak F. Involvement of the posterior tool processing network during explicit retrieval of action tool and semantic tool knowledge: an fMRI study. Cereb Cortex. 2023 May 24;33(11):6526-6542. doi: 10.1093/cercor/bhac522. PMID 36721902
- [Background] Federico G, Cavaliere C, Reynaud E, Salvatore M, Brandimonte MA, Osiurak F. The Area Prostriata may play a role in technical reasoning. Behav Brain Funct. 2022 Nov 25;18(1):12. doi: 10.1186/s12993-022-00200-9. PMID 36434696
- [Background] Federico G, Reynaud E, Navarro J, Lesourd M, Gaujoux V, Lamberton F, Ibarrola D, Cavaliere C, Alfano V, Aiello M, Salvatore M, Seguin P, Schnebelen D, Brandimonte MA, Rossetti Y, Osiurak F. The cortical thickness of the area PF of the left inferior parietal cortex mediates technical-reasoning skills. Sci Rep. 2022 Jul 12;12(1):11840. doi: 10.1038/s41598-022-15587-8. PMID 35821259